CLINICAL TRIAL: NCT03145623
Title: Retrospective Efficacy and Safety Study With Elbasvir 50 mg/Grazoprevir 100 mg in HCV-infected Patients With Chronic Kidney Disease Stage 4-5 During the French Temporary Authorization for Use (ATU) Program: Data From Real-life
Brief Title: Retrospective Efficacy and Safety Study With Elbasvir/Grazoprevir in HCV-infected Patients With Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Collaborators: MSD France (Industry)
Responsible Party: Sponsor
Other Study IDs: RC31/17/0096
Record Dates: First submitted 2017-04-25; First posted 2017-05-09 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Hepatitis C; Chronic Kidney Diseases
MeSH Terms: conditions — Hepatitis C; Renal Insufficiency, Chronic | interventions — elbasvir-grazoprevir drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Elbasvir and Grazoprevir — Elbasvir 50 mg and grazoprevir 100 mg during the French temporary authorization for use (ATU) program

SUMMARY:
Retrospective Efficacy and Safety Study With Elbasvir (EBR) 50 mg/Grazoprevir (GZR) 100 mg in Hepatitis C Virus (HCV)-infected Patients With Chronic Kidney Disease (CKD) Stage 4-5 During the French Temporary Authorization for Use (ATU) Program: Data From Real-life

DETAILED DESCRIPTION:
Primary objective : Retrospectively collect and describe the real life efficacy (SVR 12)* and safety data of EBR 50 mg/GZR 100 mg based therapy, 12 or 16 weeks dosed in HCV-infected patients with chronic kidney disease. These data are collected following French ATU allocation.

ELIGIBILITY:
Inclusion Criteria:

* documented chronic (at least 6 months) HCV Genotype1 (GT1) and Genotype 4 (GT4) infection
* Mono infected by HCV or co-infected by HCV and HIV
* Have an HCV treatment status corresponding to one of the following:

  1. Treatment-naïve: Naïve to all anti-HCV treatment
  2. Prior interferon or pegylated interferon + ribavirin treatment failure (null responders, partial responders, relapsers)
  3. Prior Interferon (IFN) or pegylated (PEG)-IFN + ribavirin + telaprevir or boceprevir or simeprevir treatment failures
  4. Prior sofosbuvir based therapy failures
  5. Pegylated interferon ribavirin intolerant
* Have CKD defined as:

Subjects with glomerular filtration rate (GFR) ≤30 ml/min who are non-dialysis dependent (NDD) or have been on hemodialysis (HD) for at least 3 months (including subjects awaiting kidney transplant and subjects with failed kidney transplants no longer on immunosuppressant therapy).

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CKD subjects with GT1 and GT4 HCV, compensated cirrhotic or non-cirrhotic (i.e all subjects with EBR 50 mg/GZR 100 mg based therapy in ATU allocation) will be included in this retrospective analysis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Efficacy of Elbasvir (EBR)/Grazoprevir (GZR) | 12 weeks after the end of all study therapy
  Describe the real life efficacy (Sustained Virologic Response SVR 12) of EBR 50 mg/GZR 100 mg based therapy by assessment of the HCV RNA

SECONDARY OUTCOMES:
Safety during treatment | during treatment
  Assessment of all Adverse Events and laboratory tests collected during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Laurent ALRIC, MD, Principal Investigator — University Hospital, Toulouse
Locations (2):
- France (2):
  - University Hospital, Caen
  - University Hospital Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No